CLINICAL TRIAL: NCT05164146
Title: The Comparison of Hypotension Incidence Between Remimazolam and Propofol in Hypertensive Patients Undergoing Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2021-1456
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Patients Undergoing Neurosurgery
MeSH Terms: interventions — Propofol; remimazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Active Comparator): During the induction, propofol was controlled according to sedline (Psi target 40)
  Interventions: Drug: propofol
- remimazolam group (Experimental): During induction, remimazolam dose was controlled according to sedline (Psi target 40)
  Interventions: Drug: remimazolam

INTERVENTIONS:
Drug: propofol — during the induction, remimazolam dose was controlled according to sedline (Psi target 40)
  Arms: propofol group
Drug: remimazolam — During induction, remimazolam dose was controlled according to sedline (Psi target 40)
  Arms: remimazolam group

SUMMARY:
This study aims to find an excellent drug in terms of hemodynamic stability when comparing the propofol and remifentanil with the combined use of remimazolam and remifentanil. When the mean blood pressure falls by 20% or more from the baseline mean blood pressure, it is considered hypotension, and a vasopressor such as ephedrine, phenylephrine, or norpin is used to control the blood pressure to within 20% of the baseline blood pressure. If the blood pressure increases by 20% or more above the baseline mean blood pressure, nicardipine infusion or remimazolam, propofol or remifentanil should be increased to control the blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. hypertension
2. patients undergoing neurosurgery
3. ASA I-III
4. 19-75 year-old patients

Exclusion Criteria:

1. emergency
2. Patients admitted on the day of surgery
3. cardiac disease
4. liver failure or liver cirrhosis
5. increased intracranial pressure(IICP)
6. mental change
7. Foreigner
8. iliteracy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
incidence of hypotension events | procedure (during induction before the surgery)
  Hypotension is considered when the mean blood pressure is 20% or more below the baseline mean blood pressure.

SECONDARY OUTCOMES:
blood pressure | procedure (during induction before the surgery)
  Blood pressure will be recorded from the start of drugs infusion to 10 minutes after intubation every 1 minutes, and they will be compared between two groups.
heart rate | procedure (during induction before the surgery)
  heart rate will be recorded from the start of drugs infusion to 10 minutes after intubation every 1 minutes, and they will be compared between two groups.
sedline psi | procedure (during induction before the surgery)
  sedline psi will be recorded from the start of drugs infusion to 10 minutes after intubation every 1 minutes, and they will be compared between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sujung Park, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi SH, Min KT, Park EK, Park S. Comparison of hypotension incidence between remimazolam and propofol in patients with hypertension undergoing neurosurgery: prospective, randomized, single-blind trial. BMC Anesthesiol. 2024 Jun 4;24(1):198. doi: 10.1186/s12871-024-02578-7. PMID 38834996